CLINICAL TRIAL: NCT01437917
Title: NOMAC : New Tools for Managing the Fate of Cereal Nutrients in the Gut : Effects of Amylose Content on Glycemic Index.
Acronym: NOMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: LOC/11-05 - NOMAC; 2011-A00517-34 (Other: ID RCB); 11/19-808 (Other: CPP Ouest V); B110607-50 (Other: AFSSAPS)
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: glycemic index
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bread with 20% amylose content (Experimental): Bread with 20% amylose content
  Interventions: Other: 20% amylose bread
- Bread with 10% amylose content (Experimental): Bread with 10% amylose content
  Interventions: Dietary Supplement: 10% amylose bread
- carbohydrates (Experimental): 50g of carbohydrates ingested with 400 ml of water
  Interventions: Dietary Supplement: Carbohydrates

INTERVENTIONS:
Other: 20% amylose bread — 20% amylose bread
  Arms: Bread with 20% amylose content
Dietary Supplement: 10% amylose bread — 10% amylose bread
  Arms: Bread with 10% amylose content
Dietary Supplement: Carbohydrates — 50g of carbohydrates ingested with 400 ml of water
  Arms: carbohydrates

SUMMARY:
The consumption of cereals-based foods with low glycemic indexes, high micronutrients and fibers contents are highly recommended. The target of this work is to provide new solutions for cereal based foods: the knowledge and understanding on the in vivo fate will be used to define structural features to gain in foods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual,
* Age between 19-65 years
* With normal food habits with at least 2 main meals per day
* Non smoking
* Having filled the consent form

Exclusion Criteria:

* BMI > 25 kg/m2,
* Diabetes or any illness susceptible to alter
* Coeliac disease
* Past history of intestinal diseases.
* Treatment susceptible of modifying glycemia.
* Allergy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Glycemic index for each bread | 2 hours
  To compare the glycemic index of breads made with different amylose content. (S1 to S6) A total of 6 visits. In each visit, blood samples will be taken for measurement of glycemia and insulinemia over 2 hours after ingestion of 50 of carbohydrates ingested with 400 ml of water.

SECONDARY OUTCOMES:
AUC for insulinemia for the 2 hours following the ingestion of each bread. | 2 hours
  To compare the AUC for insulinemia for the 2 hours following the ingestion of each bread.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BONNET, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France